CLINICAL TRIAL: NCT00290069
Title: Comparative Study of Tacrolimus and Rapamycin to Evaluate the Renal Function in Patients Older Than 50 Years, Receptors of a Kidney From a Donor Older Than 55 Years in a Mycophenolate Mofetil and Daclizumab Immunosuppressor Regime
Brief Title: Renal Function Optimization With Mycophenolate Mofetil (MMF) Immunosuppressor Regimes (ALHAMBRA)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sociedad Andaluza de Trasplantes de Organos y Tejidos (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SATOT42005; EudraCT number: 2005-001854-25; ALHAMBRA
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2006-02

CONDITIONS: Kidney Diseases; Graft Rejection
Keywords: Renal function; Serum creatinine; Immunosuppression; Rejection
MeSH Terms: conditions — Kidney Diseases; Rejection, Psychology | interventions — Tacrolimus; Sirolimus

INTERVENTIONS:
Drug: Tacrolimus
Drug: Rapamycin

SUMMARY:
The main aim of this study is to compare the renal function (serum creatinine at 6 months) in the later introduction of tacrolimus or rapamycin based in immunosuppressor regimes with daclizumab, mycophenolate mofetil, and steroids in patients older than 50 years of age who are the recipients of a graft from donors aged 55 years and older.

DETAILED DESCRIPTION:
The study population characteristics raise the need to establish a treatment regime that assures suitable intensity immunosuppression to avoid the appearance of rejection episodes, but minimizes the doses to prevent over-immunosuppression in a population with a theoretic minor immune response.

On the other hand, the delay in the introduction of calcineurin inhibitors will prevent increasing the risk of early graft dysfunction allowing the highest post-transplant renal recovery in organs with less operative mass and greater sensibility to the nephrotoxic effect of these drugs.

The results of several studies confirm the goodness of regimes that include low doses of calcineurin inhibitors, delay their introduction or avoid them.

Nevertheless, although it is standard practice to evaluate the effectiveness of the regimes for a time to assure, with certainty, the response to the treatments, these follow-ups are still relatively short to assure the efficacy for a long-term study and to detect the problems. The studies with a high number of patients and long follow-up periods are difficult, so several authors have proposed different alternatives of control in a short-term study that could be useful as surrogate markers or predictive efficacy variables for the long term.

If the drug or study regime is efficient, the observed change after the transplantation surgery will have to be fast and objective. The increase of serum creatinine between 6 and 12 months post-transplant is a reliable marker of graft failure risk, and the magnitude of the serum creatinine change in these months is a marker of the relationship with long-term survival. For that reason, renal function (serum creatinine) is included as a main efficacy variable.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients older than 50 years who are primary recipients of a renal allograft from a donor older than 55 years.
* Patients who have given their consent previously to their participation in the study.

Exclusion Criteria:

* Recipients of a multi-organ transplant.
* Recipients of a transplant from a cadaveric donor with a cold ischemic time > 30 hours.
* Patients with a plasma renin activity (PRA) > 20% in 6 months previous to the inclusion.
* Breast-feeding, pregnant, or fertile women who do not use a reliable anticonceptive method before starting therapy with the study drug, during the therapy, and during the 4 months after the last dose of the drugs administered in the study.
* Patients with leukocyte count < 2.5 x 10^9/L, platelet count < 100 x 10^9/L, or haemoglobin < 6 g/dL in the inclusion time
* Patients with active hepatic illness evidence.
* Patients with active peptic ulcer.
* Patients with serious diarrhoea or any intestinal upset that may interfere in the absorption capability of oral medication, including diabetic patients with previously diagnosticated diabetic gastroenteropathy.
* Patients with evidence of active systemic infection that require the continued use of antibiotics or evidence of HIV infection or hepatitis B presence (positive HBs-Ag) or active chronic hepatitis C.
* Patients with malignancy history (except satisfactorily treated non- melanocytic localized skin cancer and cervix "in situ" carcinoma).
* Patients with history of psychologic disease that may interfere in the patients capability to understand the study requirements.
* Patients who the investigator thinks need a treatment with any medication listed below:

  * Azathioprine,
  * Methotrexate,
  * Cyclofosfamide,
  * Polyclonal or monoclonal anti-lymphocitaries antibodies (OKT3, ATG), used for the induction in patients with high immunologic risk,
  * Basiliximab, and
  * Other research drugs
* Known hypersensibility or complete contraindication of any of the drugs administered in the study context or any other substance present in the study drugs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine at 6 months

SECONDARY OUTCOMES:
Calculated creatinine clearance (Cockroft Gault)
Acute rejection rate at 6 months and time until first rejection
Patient and graft survival at 6 months
Rate and length of the delay in the graft function defined as dialysis in the first week post-transplant
Treatment failure at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Gonzalez Molina, MD, Principal Investigator — Sociedad Andaluza de Trasplantes de Organos y Tejidos
Locations (7):
- Spain (7):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario La Fe, Valencia, Valencia